CLINICAL TRIAL: NCT04941989
Title: A Phase 1, Randomised, Double-Blind, Placebo-Controlled, First in Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Subcutaneous HTL0022562 in Healthy Adult Subjects
Brief Title: A Study in Healthy Subjects to Assess the Safety, Tolerability and Pharmacokinetics of HTL0022562
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Early termination of study pending evaluation of emerging preclinical profile.
Sponsor: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HTL0022562-101; 2020-002887-30 (EudraCT Number); 246780 (Other: Parexel Early Phase Clinical Unit London)
Record Dates: First submitted 2021-06-08; First posted 2021-06-28 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: First in Human; Single Ascending Dose; Multiple Ascending Dose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 Single Ascending Dose (Experimental): Eight subjects in up to 7 cohorts will be dosed. One or more subcutaneous injections of HTL0022562 will be administered. In each cohort, 6 subjects will receive HTL0022562 and 2 subjects will receive placebo.
  Interventions: Drug: HTL0022562; Drug: Placebo
- Part 2 Multiple Ascending Dose (Experimental): Eight subjects in up to 4 cohorts will be dosed, following safety, tolerability and pharmacokinetic (PK) review of completed dose of Single Ascending Dose Cohort 5. In each cohort, 6 subjects will receive HTL0022562 and 2 subjects will receive placebo.
  Interventions: Drug: HTL0022562; Drug: Placebo

INTERVENTIONS:
Drug: HTL0022562 — HTL0022562
Drug: Placebo — Placebo

SUMMARY:
Phase 1, randomised, double-blind, first in human, two part, single centre, placebo controlled, single and multiple ascending dose trial in healthy adult subjects to evaluate the safety, tolerability and pharmacokinetics of HTL0022562.

DETAILED DESCRIPTION:
This is a first in human, two part, double blind, placebo controlled, randomised single and multiple ascending subcutaneous dose study to evaluate the safety, tolerability and pharmacokinetics of HTL0022562.

Part 1 comprises of 7 sequential ascending dosing cohorts and Part 2 comprises of 4 multiple ascending dosing cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males or healthy females of non-childbearing potential (WoNCBP) aged 18 to 55 years inclusive, with a body mass index >18.5-<30kgm2 and body weight ≥50kg.
* Healthy on the basis of a clinical history, physical examination, electrocardiogram (ECG), vital signs and laboratory tests of blood and urine.
* Willingness to comply with requirements or the trial, including contraception requirements.
* Able to give fully informed consent.

Key Exclusion Criteria:

* Confirmed current Coronavirus Disease 2019 (COVID 19) infection before randomisation.
* Clinical signs and symptoms consistent with COVID 19 (e.g. fever, dry cough, dyspnoea, sore throat, or fatigue) or confirmed infection by appropriate laboratory test within the last 4 weeks prior to Screening or on admission.
* Suffered from severe course of COVID 19 (extracorporeal membrane oxygenation (ECMO), mechanically ventilated).
* Receipt of any investigational medicinal product (IMP) in a clinical research study within the previous 3 months (or 5 half-lives, whichever is longer) of Screening.
* Any abnormalities on 12-lead ECG or BP at Screening (as specified).
* History of any drug or alcohol abuse in the past 2 years.
* Vital signs outside the normal range for healthy volunteers
* Clinically significant abnormal biochemistry, haematology, coagulation, or urinalysis
* Abnormal renal function, hepatic function or history of abnormal hepatic function occurring during treatment with investigational or licensed drugs, which led to permanent discontinuation of treatment.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti HCV), or human immunodeficiency virus (HIV)
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, or current hepatic renal dysfunction as judged by the investigator.
* Risk factor for ischaemic heart disease or cerebrovascular disease.
* Failure to satisfy, in the Investigator's judgement, the subject's fitness to participate for any other reason, including previous serious adverse reaction or serious hypersensitivity reactions to any drug or formulation excipients administered parenterally or orally.
* All female subjects must have a negative serum and urine pregnancy test at Screening and admission, respectively.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) | Screening up to post last dose: Day 8 (Part 1) / Day 15 (Part 2)
  All Adverse Events (AEs), including clinical laboratory, vitals signs, body temperature, respiratory rate, physical examinations, local tolerability and site injection reactions, and ECGs will be analyzed in all subjects.

SECONDARY OUTCOMES:
Part 1 and Part 2: Cmax | Part 1 up to Day 8, Part 2 up to Day 15
  Plasma pharmacokinetic parameter: maximum systemic concentration of HTL0022562
Part 1 and Part 2: Tmax | Part 1 up to Day 8, Part 2 up to Day 15
  Plasma pharmacokinetic parameter: time to Cmax of HTL0022562
  Plasma pharmacokinetic parameter: time to Cmax of HTL0022562
Part 1 and Part 2: Area Under Curve (AUC) | Part 1 up to Day 8, Part 2 up to Day 15
  Plasma pharmacokinetic parameter: Area under the plasma concentration versus time curve derived from systemic concentrations of HTL0022562
Part 1 and Part 2: Ae | Part 1 up to Day 8, Part 2 up to Day 15
  Urine pharmacokinetic parameter: Amount of HTL0022562 recovered in urine for each urine collection interval

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel Early Phase Clinical Unit, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No